CLINICAL TRIAL: NCT01951846
Title: An Open Label Dose Escalation Study of BIBF 1120 Administered Orally for Four Weeks in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: To Determine the Maximum Tolerated Dose (MTD) of BIBF 1120 in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 1199.1
Record Dates: First submitted 2013-09-17; First posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Malignant Solid Tumour
MeSH Terms: interventions — nintedanib

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120

SUMMARY:
The primary objective of this study was to determine the maximum tolerated dose (MTD) of BIBF 1120 in patients with solid tumours by the monitoring of drug-related adverse events. Secondary objectives were the evaluation of safety, efficacy, pharmacokinetics, and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumours, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
* Evaluable tumour deposits by one or more techniques (X-ray, CT, MRI, ultrasound)
* Age 18 years or older
* Life expectancy of at least three months
* Patients had to give written informed consent (which must be consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) and local legislation)
* Eastern Cooperative Oncology Group (ECOG) performance score < 2
* Full recovery from all therapy-related toxicities from previous chemo-, hormone-,immuno-, or radiotherapy

Exclusion Criteria:

* History of relevant surgical procedures during the last four weeks prior to treatment with the trial drug, or active ulcers, or injuries with incomplete wound healing
* Pregnancy or breastfeeding
* Active infectious disease
* Brain metastases requiring therapy
* Absolute neutrophil count less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin greater than 1.5 mg / dl (> 26 μmol / L, International System of Units (SI unit) equivalent)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg / dl (> 132 μmol / L, SI unit equivalent)
* Uncontrolled, severe hypertension
* Gastrointestinal disorders anticipated to interfere with the resorption of the study drug
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-11; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of BIBF 1120 | up to 30 days

SECONDARY OUTCOMES:
Overall best investigator assessment of tumour response | up to 4 months
Overall best calculated assessment of tumour response | up to 4 months
Time to tumour progression | up to 4 months
Change in Eastern Cooperative Oncology Group (ECOG) score | up to 4 months
Number of patients with response in transfer of contrast medium into tissue (Ktrans) | up to 4 months
Number of patients with response in initial area under the curve for first 60 seconds after onset of gadolinium uptake (iAUC60) | 60 seconds
Mean plasma level of vascular endothelial growth factor (VEGF) | 10 hours after drug intake
Mean plasma level of basic fibroblast growth factor (bFGF) | 10 hours after drug intake

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Tumorbiologie, Abteilung Internistische Onkologie, Freiburg im Breisgau, Germany